CLINICAL TRIAL: NCT05825560
Title: Opioid-free Analgesia in Intensive Care Unit: a Prospective, Monocentric, Randomized, Double Blind, Feasability Clinical Trial
Brief Title: Opioid-free Analgesia in Intensive Care Unit
Acronym: OFICU
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LOCAL/2022/RW-01; 2022-003273-37 (EudraCT Number)
Record Dates: First submitted 2023-04-11; First posted 2023-04-24 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Intubation
Keywords: orotracheal intubation; mechanical ventilation; sedation analgesia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Analgesia combines paracetamol (1g every 6 to 8 hours according to age and weight recommendations) and remifentanil, adapted according to a tiered administration system depending on the Behavior Pain Scale (BPS) and the theoretical ideal weight. Remifentanil doses are adjusted so that the patient has a BPS score of 4 or less. Reassessment of analgesia will be carried out every 30 minutes until analgesic adaptation is complete, then every 2 hours as is usually done in our department.
  If the BPS is less than or equal to 4, the therapeutic de-escalation will be done with a reverse algorithm until the analgesic drugs are stopped.
  After the sedation balance phase, the patient's BPS will be assessed every 2 hours.
  Interventions: Drug: Standard multimodal analgesia
- OFA Group (Experimental): A fixed combination of nefopam and tramadol will be initiated at daily doses. An initial dose of 50mg tramadol and 20mg nefopam IV over 30 min. will be administered. Reassessment of analgesia will be performed every 30 min. for two hour and then every 2 hours.
  * If BPS is > 4, administration of ketamine with an initial bolus of 0.15mg/kg followed by continuous administration at a dose of 0.15mg/kg/hour.
  * If the BPS is < 4, remifentanil is introduced at the minimum effective dose, in a stepwise fashion according to the theoretical ideal weight
  * In the event of maximum pain requiring the full range of therapies in the algorithm the total dose of tramadol will be 450mg/day and nefopam 120mg/day, in accordance with summaries of product characteristics.
  * If the BPS < or = 4, the therapeutic de-escalation will be done with a reverse algorithm until the analgesic drugs are stopped, according to the following scheme: remifentanil, ketamine, tramadol and then nefopam.
  Interventions: Drug: OFA multimodal analgesia

INTERVENTIONS:
Drug: OFA multimodal analgesia — Multimodal opioid free analgesia
  Arms: OFA Group
Drug: Standard multimodal analgesia — Standard remifentanil analgesia
  Arms: Control group

SUMMARY:
ICU patients experience moderate to severe pain. Studies and guidelines point out the benefits of multimodal analgesia on pain control, opioid spare and on lowering its adverse effects. However, no recommendation about drugs or protocol has been formulated. In our study, investigators studied the feasibility and the impact on Remifentanil spare of a standardized protocol using multimodal analgesia (Paracetamol, Nefopam, Tramadol, Ketamine, Remifentanil) compared to the standard-of-care strategy using Paracetamol and Remifentanil. The investigators conducted a prospective, ''proof of concept'', randomized, double-blind, parallel group, placebo-controlled trial. The investigators studied multimodal analgesia versus standard-of-care in ICU patients requiring sedation-analgesia for invasive mechanical ventilation.The investigators hypothesized that Remifentanil consumption decrease by 15% with the use of a standardized multimodal analgesia strategy

DETAILED DESCRIPTION:
ICU patients requiring sedation-analgesia for mechanical ventilation for at least 48 hours are randomized in 2 parallel groups : control arm using ''standard of care'' analgesia (Paracetamol and Remifentanil), and interventional arm using multimodal analgesia at different level according to pain accessed by BPS (Step 1 : Paracetamol, Nefopam, Tramadol, Step 2 : Ketamine, Step 3 : Remifentanil). Sedation drugs are standard of care (Propofol and Midazolam if Propofol isn't enough) to obtain prescribed sedation accessed by RASS. Double-bling is kept for 72 hours until the primary outcome is obtained.

The investigators hypothesize a 15% reduction of Remifentanil consumption in the interventional group.

ELIGIBILITY:
Inclusion Criteria:

* Patient hospitalized in ICU and requiring sedation-analgesia for mechanical ventilation.
* Patient undergoing mechanical ventilation for more than 2 hours and less than 24 hours.
* Informed consent signed by the patient or his trusted person, legal representative, family member, curator or tutor, or emergency consent procedure.
* Patient affiliated to the French Government Public Health Insurance.
* Patient over 18 years old.

Exclusion Criteria:

* Patient already involved in a trial that might influence our primary endpoint.
* Patient in exclusion-period determined by another trial or study.
* Patient who is likely to be requiring less than 48 hours of mechanical ventilation.
* Patient with contraindication or allergies to at least one of the following medication : paracetamol, nefopam, tramadol, ketamine, remifentanil.
* Patient with hepatic insufficiency (defined as PT < 50%).
* Parturient or breast-feeding patient.
* Patient suffering from moderate to severe Acute Respiratory Distress Syndrome (ARDS), with decreased PaO2/FiO2 ratio under 150mmHg after respiratory optimization (courant volume 6mL/kg and PEEP > 5mbar).
* Patient requiring curare treatment.
* Patients with an indication for locoregional analgesia prior to extubation (perineural sealing, epidural analgesia).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
Daily remifentanil consumption (after randomisation) | 48th hour after randomisation
  daily consumption of remifentanil between the 24th hour and the 48th hour after randomisation of patients admitted to the ICU and requiring at least 48 hours of mechanical ventilation

SECONDARY OUTCOMES:
Impact of a non-opioid analgesia strategy on morphine savings at D7 | Day 28
  Cumulative dose of remifentanil
Impact of an opioid-free analgesia strategy on sedative consumption | Day 28
  Number of lived days free of remifentanil
Impact of an opioid-free analgesia strategy on sedative consumption | Day 28
  Daily consumption of sedative drugs from inclusion to D28
Impact of a non-opioid analgesia strategy on the duration of mechanical ventilation | Day 28
  Number of live days free of mechanical ventilation
Impact of an opioid-free analgesia strategy on norepinephrine | Day 28
  Number of lived days free of norepinephrine
Impact of a non-opioid analgesia strategy on organ failure at D28 | Day 28
  SOFA Score (Sepsis-related Organ Failure Assessment)
Impact of a non-opioid analgesia strategy on fluid intake | Day 28
  Daily fuid intake in milliliter
Impact of a non-opioid analgesia strategy on mental confusion | Day 28
  CAM ICU test
Impact of a non-opioid analgesia strategy on the occurrence of morphine-related adverse events | Day 28
  Presence of one or more events of special interest or expected adverse events: constipation, bradycardia, bladder globe, nausea, vomiting, liver disturbance, serotonin syndrome
Impact of a non-opioid analgesia strategy on the incidence of ventilator-associated pneumonia | Day 28
  Presence of pneumonia associated with mechanical ventilation
Impact of a non-opioid analgesia strategy on extubation failure rates | 48 hours after extubation
  extubation failure and cause (reintubation within 48 hours of first extubation)
Impact of a non-opioid analgesia strategy onICU and hospital length of stay | Day 90
  Length of stay in the intensive care unit and in the hospital
Impact of the non-opioid analgesia strategy on vital prognosis at D28 and D90. | Day 90
  Vital status at day 28 and day 90
Impact of a non-opioid analgesia strategy on morphine dependence at D90 | Day 90
  Opioid use at D90

CONTACTS AND LOCATIONS:
Locations (1):
- Remy WIDEHEM, Nîmes, Gard, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wheeler KE, Grilli R, Centofanti JE, Martin J, Gelinas C, Szumita PM, Devlin JW, Chanques G, Alhazzani W, Skrobik Y, Kho ME, Nunnally ME, Gagarine A, Ergan BA, Fernando S, Price C, Lewin J, Rochwerg B. Adjuvant Analgesic Use in the Critically Ill: A Systematic Review and Meta-Analysis. Crit Care Explor. 2020 Jul 6;2(7):e0157. doi: 10.1097/CCE.0000000000000157. eCollection 2020 Jul. PMID 32696016
- [Background] Devlin JW, Skrobik Y, Gelinas C, Needham DM, Slooter AJC, Pandharipande PP, Watson PL, Weinhouse GL, Nunnally ME, Rochwerg B, Balas MC, van den Boogaard M, Bosma KJ, Brummel NE, Chanques G, Denehy L, Drouot X, Fraser GL, Harris JE, Joffe AM, Kho ME, Kress JP, Lanphere JA, McKinley S, Neufeld KJ, Pisani MA, Payen JF, Pun BT, Puntillo KA, Riker RR, Robinson BRH, Shehabi Y, Szumita PM, Winkelman C, Centofanti JE, Price C, Nikayin S, Misak CJ, Flood PD, Kiedrowski K, Alhazzani W. Clinical Practice Guidelines for the Prevention and Management of Pain, Agitation/Sedation, Delirium, Immobility, and Sleep Disruption in Adult Patients in the ICU. Crit Care Med. 2018 Sep;46(9):e825-e873. doi: 10.1097/CCM.0000000000003299. PMID 30113379
- [Derived] Widehem R, Nicolet C, Delannoy V, Barthelemi L, Soulairol I, Lefrant JY, Mura T, Roger C. Effect of a multimodal analgesia strategy on remifentanil daily consumption in mechanically ventilated adult ICU patients: study protocol for a randomised, placebo-controlled, double-blind, parallel-group clinical trial. BMJ Open. 2025 Jan 20;15(1):e090396. doi: 10.1136/bmjopen-2024-090396. PMID 39832962